CLINICAL TRIAL: NCT05467566
Title: The Effects of Transcranial Direct Current Stimulation Combined With Pilates Based Exercise in the Treatment of Patients With Chronic Low Back Pain
Brief Title: Transcranial Direct Current Stimulation Combined With Exercise in Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Liane de Brito Macedo, Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LBPETCC22
Record Dates: First submitted 2022-07-15; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Low Back Pain; Transcranial Direct Current Stimulation
Keywords: Transcranial Direct Current Stimulation; Low back pain; Exercise; Chronic pain; Combined modality therapy; Motor cortex
MeSH Terms: conditions — Low Back Pain; Motor Activity; Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation + exercise group (Experimental): 30-minute exercise program (based on Pilates method) combined with active transcranial direct current stimulation.
  Interventions: Device: Transcranial direct current stimulation
- Sham stimulation + exercise group (Sham Comparator): This arm will perform the same procedures of experimental group but the stimulator will be turned off after 30 seconds and the volunteers will not receive current for the rest of the session.
  Interventions: Device: Sham Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Exercise protocol + application of active direct current stimulation for 30 minutes.
  Arms: Stimulation + exercise group
Device: Sham Transcranial direct current stimulation — Exercise protocol + application of simulation of direct current stimulation for 30 minutes. The stimulator will be turned off after 30 seconds and the volunteers will not receive current for the rest of the session.
  Arms: Sham stimulation + exercise group

SUMMARY:
The purpose of this study is to evaluate the effects of transcranial direct current stimulation combined with Pilates based exercise on chronic low back pain. This is a randomized clinical trial composed of two arms.

DETAILED DESCRIPTION:
Chronic low back pain may be associated with pathoanatomical, neurophysiological, physical, psychological and social factors. Treatments that relieve the symptoms of these patients are of great importance to improve the quality of life of these individuals. Thus, this study aims to evaluate the effects of transcranial direct current stimulation combined with Pilates based exercise on chronic low back pain. This is a randomized clinical trial that will be composed of men and women between 18 and 65 years of age, with a history of low back pain for more than 12 weeks and a minimum pain intensity equal to 3 cm on the numerical pain scale. The volunteers will be randomized into two distinct groups: stimulation + exercise group (EG - will perform a Pilates based exercise protocol combined with transcranial direct current stimulation) and sham stimulation + exercise group (SG - will perform the same exercise program combined with sham stimulation). The interventions, regardless of the group, will be carried out three times a week for four weeks. Participants will be submitted to three assessments: the first (T0) will be performed before the treatment protocols; the second (T1) will be performed after the four weeks of intervention; and the third (T2) will be a follow-up one month after the end of the treatment protocol. Pain sensation, functional performance, central sensitization, quality of life, pressure pain threshold, global impression of change, adverse events and medication use will be evaluated. For the statistical analysis, a mixed model ANOVA will be performed for the inter and intragroup comparison, with Tukey's post hoc, considering a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with chronic nonspecific low back pain (for more than 12 weeks) and minimum pain intensity of 3 on numerical pain rating scale.

Exclusion Criteria:

* diagnosis of fracture and spine pathologies, fibromyalgia, spine surgery in the last year;
* low cognitive level assessed by the Mini Mental State Examination;
* presence of central neurological diseases (such as Parkinson's and stroke) or psychiatric (such as depression or schizophrenia);
* history of epileptic illness;
* seizure history;
* brain implants;
* pacemaker;
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Change from baseline in pain intensity at four weeks after intervention and 1 month of follow-up
  Pain intensity measured by numerical pain rating scale (11 points scale)
Functional performance associated to back pain | Change from baseline in functional performance at four weeks after intervention and 1 month of follow-up
  Functional performance associated with low back pain measured by Roland Morris Disability Questionnaire (24 itens)

SECONDARY OUTCOMES:
Pressure pain threshold | Change from baseline in pressure pain threshold at four weeks after intervention and 1 month of follow-up
  Pressure pain threshold measured by pressure algometer.
Individual quality of life | Change from baseline in quality of life questionnaires at four weeks after intervention and 1 month of follow-up
  Measurement of quality of life using SF-36 questionnaire (36 items, divided into 8 subscales)
Patient global impression of change | Change from baseline in Patient global impression of change at each intervention day and at four weeks of intervention and 1 month of follow-up.
  Patient global impression of change measured by a scale with seven points, where 1 is equal to no change or worse and 7 is much better.
Central Sensitization | Change from baseline of central sensitization at four weeks after intervention and 1 month of follow-up.
  Evaluation of Central Sensitization using Central Sensitization Inventory (CSI).The questionnaire is divided into two parts, the first with a score from 0 to 100 measures 25 somatic and emotional symptoms, while the second part relates to specific previous diagnoses.
Adverse events | Up to 4 weeks of intervention and 1 month of follow-up.
  Patient perception of any adverse event during the intervention protocol.
Use of medications | Up to 4 weeks of intervention and 1 month of follow-up.
  Patient declaration of medication use.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] da Silva AAC, Gomes SRA, do Nascimento RM, Fonseca AK, Pegado R, Souza CG, Macedo LB. Effects of transcranial direct current stimulation combined with Pilates-based exercises in the treatment of chronic low back pain in outpatient rehabilitation service in Brazil: double-blind randomised controlled trial protocol. BMJ Open. 2023 Dec 30;13(12):e075373. doi: 10.1136/bmjopen-2023-075373. PMID 38159941